CLINICAL TRIAL: NCT01579708
Title: Evaluation of the Program SI! for Preschool Education: A School-Based Randomized Controlled Trial
Acronym: Preschool_PSI!
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fundación Centro Nacional de Investigaciones Cardiovasculares Carlos III (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Preschool_PSI!
Record Dates: First submitted 2012-04-16; First posted 2012-04-18 (Estimated); Last update posted 2017-12-21 (Actual); Status verified 2017-12

CONDITIONS: Healthy Lifestyle; Cardiovascular Disease
Keywords: Diet; Physical activity; Knowledge; Attitudes; Habits; Lifestyle; School-based
MeSH Terms: conditions — Cardiovascular Diseases; Motor Activity; Behavior; Habits

ARMS (2):
- Program SI! educational intervention (Experimental)
  Interventions: Behavioral: Program SI! educational intervention
- Control (No Intervention)

INTERVENTIONS:
Behavioral: Program SI! educational intervention — School-based educational program to improve the knowledge, the attitudes, and the habits of children, their parents and teachers, with respect to a healthy lifestyle behavior.
  Arms: Program SI! educational intervention

SUMMARY:
Cardiovascular disease continues to be the principal cause of death in the world. At present, the risk factors for cardiovascular disease continue to appear at an earlier age permitting prevention activities and the promotion of healthy habits to focus on children. Numerous studies have shown that these factors can be controlled in children through school-based interventions. At the same time, data shows that there is a persistence of unhealthy lifestyles (ie sedentary lifestyles, the use of tobacco, etc…) that begin in childhood and are perpetuated until adulthood. Therefore, the acquisition of healthy lifestyles should begin as early as possible. The SI Program for Preschool Education is an intervention that is both school and home based designed to improve the habits, knowledge and attitudes in four key areas: Food (diet), Physical Activity, Knowledge of the Body and Managing Emotions. This intervention will be implemented in children from three to five years of age, in their parents and in their teachers. To evaluate the efficacy of this intervention, the principal aim of the phase of evaluations is to quantify the behavior changes in the three groups/populations mentioned. The evaluation has been designed according to the controlled intervention model, in which twenty-four schools from the Community of Madrid will be randomized to implement the Program si! for Preschool Education or to function as control schools.

ELIGIBILITY:
Inclusion Criteria:

* The schools must be located within the municipality of Madrid
* The schools must be public
* The schools must have, at the least, two classes for Preschool Education, for children 3, 4 and 5 years of age
* The schools must make available the use of the cafeteria.

Exclusion Criteria:

* NA

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2060 (Actual)
Dates: Start 2011-09; Primary Completion 2012-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
1-year, and 3-year changes from baseline in questionaires scores for knowledge, attitudes, and habits of children, parents and teachers in regards to a healthy lifestyle. | 3 years

SECONDARY OUTCOMES:
1-year, and 3-year changes from baseline in body composition, and blood pressure of children. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Rodrigo Fernandez-Jimenez, MD PhD, Principal Investigator — Fundacion Centro Nacional de Investigaciones Cardiovasculares; Valentin Fuster, MD, PhD, Study Chair — Fundacion Centro Nacional de Investigaciones Cardiovasculares
Locations (1):
- Fundacion Centro Nacional de Investigaciones Cardiovasculares, Madrid, Spain

REFERENCES:
- [Derived] Penalvo JL, Santos-Beneit G, Sotos-Prieto M, Bodega P, Oliva B, Orrit X, Rodriguez C, Fernandez-Alvira JM, Redondo J, Vedanthan R, Bansilal S, Gomez E, Fuster V. The SI! Program for Cardiovascular Health Promotion in Early Childhood: A Cluster-Randomized Trial. J Am Coll Cardiol. 2015 Oct 6;66(14):1525-1534. doi: 10.1016/j.jacc.2015.08.014. PMID 26429075
- [Derived] Penalvo JL, Sotos-Prieto M, Santos-Beneit G, Pocock S, Redondo J, Fuster V. The Program SI! intervention for enhancing a healthy lifestyle in preschoolers: first results from a cluster randomized trial. BMC Public Health. 2013 Dec 20;13:1208. doi: 10.1186/1471-2458-13-1208. PMID 24359285
- [Derived] Penalvo JL, Santos-Beneit G, Sotos-Prieto M, Martinez R, Rodriguez C, Franco M, Lopez-Romero P, Pocock S, Redondo J, Fuster V. A cluster randomized trial to evaluate the efficacy of a school-based behavioral intervention for health promotion among children aged 3 to 5. BMC Public Health. 2013 Jul 15;13:656. doi: 10.1186/1471-2458-13-656. PMID 23855415
- See also: Related Info — http://www.programasi.org/